CLINICAL TRIAL: NCT05860673
Title: Minimally Invasive Surgery vs Standard Posterior Approach in the Treatment of Developmental Idiopathic Scoliosis: Randomized Trial.
Brief Title: Minimally Invasive Surgery vs Standard Posterior Approach in the Treatment of Developmental Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MISpro
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: posterior spinal fusion; mini invasive scoliosis surgery; Adolescent Idiopathic Scoliosis; randomized trial

STUDY DESIGN:
Intervention Model Description: This is a randomized trial with 1:1 allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini invasive scoliosis surgery (MIS) (Experimental): This technique involves making small, noncontiguous, midline skin incisions at the levels to be instrumented, usually proximal and distal to the area of arthrodesis. A median fascial incision is then made to expose the vertebral segments on which to thread the screws while the bar is inserted submuscularly in a cranio-caudal direction, after appropriate maneuvers to correct the deformity.
  Interventions: Procedure: mini invasive scoliosis surgery
- posterior spinal fusion technique (PSF) (Active Comparator): This technique is the surgical gold standard. It consists of an instrumented arthrodesis with posterior access and requires a wide median incision with extensive muscle dissection.
  Interventions: Procedure: posterior spinal fusion technique

INTERVENTIONS:
Procedure: mini invasive scoliosis surgery — The minimally invasive technique, involves two small median skin incisions that allow the deep structures to be exposed. The muscle fibers are separated from the bony insertion by the process of subperiosteal "skeletonization." The Investigators then proceed with the arthrectomy of the levels to be instrumented and the infiltration of pedicle screw pairs of the appropriate caliber according to the "free-hand" technique. After amplioscopic control of proper screw placement, osteotomies of the posterior elements are performed to facilitate correction of the metameres.
  Arms: mini invasive scoliosis surgery (MIS)
Procedure: posterior spinal fusion technique — The standard open technique involves a longitudinal incision along the midline extended along the entire thoracolumbar spine, the paravertebral muscles are incised and spread apart to expose the posterior vertebral structures, in a stretch extending more than 30 cm. The series of facetectomies are performed first, and then pairs of pedicle screws are infixed freehand.
  After performing the osteotomies necessary to mobilize the vertebral metameres at the apex of the deformity, correction by derotation maneuvers is continued, and the obtained correction is fixed with pre-shaped bars that are then connected to the screws and tightened to the nuts by dynamometric technique. Almost all vertebral levels of the thoracolumbar tract are included in the arthrodesis
  Arms: posterior spinal fusion technique (PSF)

SUMMARY:
This is a randomized trial with 1:1 allocation. The aim of the study is to evaluate clinical and radiographic outcomes in patients with developmental age idiopathic scoliosis treated with mini invasive scoliosis surgery (MIS) technique versus posterior spinal fusion (PSF) technique through clinical and radiographic evaluations.

DETAILED DESCRIPTION:
Patients with developmental age idiopathic scoliosis will be included in a randomized trial in which one group of patients will be treated with mini invasive scoliosis surgery technique , and one group will be treated instead with traditional posterior spinal fusion arthrodesis. The study design involves a noninferiority evaluation, assuming that MIS does not produce inferior results to the classic technique from the point of view of curve correction. This result would be important, because with equal curve correction success, the risk/benefit balance for minimally invasive surgery is superior, as it reduces the risk of transfusion and postoperative pain. The results of this study could therefore give important guidance for surgeons on choosing the optimal treatment for patients.

Patients will be evaluated by clinical examination, before the surgical procedure and at subsequent follow-ups as per clinical practice: at 2, 6, 12, 24, 60 months after treatment by medical personnel.

During the selection visit, patients will also be evaluated with radiographic examination for measurements necessary to decide the indication for surgical treatment. The patient also undergoes postoperative radiographic examination before discharge, as well as at follow-ups at 2, 6, 12, 24, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AIS
2. Age between 12 and 25 years;
3. Site of scoliotic curve: thoracic and/or lumbar;
4. Preoperative radiographic range of the main scoliotic curve between 40° and 70° according to Cobb;
5. Ability and consent of patients/parents to actively participate in the study and clinical follow-up.

Exclusion Criteria:

1. Patients already treated surgically for scoliosis;
2. Site of the scoliotic curve: cervical;
3. Patients with scoliosis other than adolescent idiopathic scoliosis;
4. Patients who do not fall within the described parameters;
5. Unbalanced sagittal profile;
6. Patients unable to consent or perform follow-ups.
7. Pregnant women.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Cobb angle measurement | 12 months follow-up
  Cobb's angle represents the gold standard for measuring the extent of the scoliotic curve; it is identified as the angle between the two lines passing through the upper limiting vertebra and the lower limiting vertebra on an antero-posterior radiogram of the spine.

SECONDARY OUTCOMES:
Cobb angle measurement | baseline (post-surgery), 2 months, 6 months, 24 months and 60 months follow-up
  Cobb's angle represents the gold standard for measuring the extent of the scoliotic curve; it is identified as the angle between the two lines passing through the upper limiting vertebra and the lower limiting vertebra on an antero-posterior radiogram of the spine.
NRS (Numeric Rating Scale) | baseline, 2 months, 6 months, 12 months, 24 months and 60 months follow-up
  NRS is a quantitative one-dimensional numerical scale, used to measure pain intensity, involves the practitioner asking the patient to select the number that best describes the intensity of his or her pain, from 0 to 10, at that specific time.
SRS-22 (Scoliosis Research Society-22) | baseline, 2 months, 6 months, 12 months, 24 months and 60 months follow-up
  SRS-22 is a questionnaire that is the most common measure for assessing quality of life in patients with spinal deformities. assesses five domains:
  1. function
  2. pain
  3. mental health
  4. self-image
  5. satisfaction/ dissatisfaction Each domain contains five questions, except for the last one, which has two questions.
  The score for each question ranges from 1 to 5. The sum of the first four domains forms an initial partial score, which can be up to 100. The total score is given by adding the last item as well, for a maximum score of 110. The purpose of the SRS-22 is to provide an assessment of pathology and patient perception regarding both the consequences of treatment choices and the effectiveness of treatment.
Oswestry Disability Index (ODI) | baseline, 2 months, 6 months, 12 months, 24 months and 60 months follow-up
  The ODI index is a valuable tool for assessing patient satisfaction in view of the patient's current clinical picture. It consists of ten sections investigating the influence of spinal pathology on different aspects of daily life: (pain intensity; personal hygiene; lifting weights; walking; sitting; standing; sleeping; sexual life; social life; traveling).
  Each section contains within it 6 possible answers with scores ranging from 0 to 5 where 0 corresponds to no difficulty or pain while 5 inability to perform the activity or disabling pain
Final treatment opinion | 2 months, 6 months, 12 months, 24 months and 60 months follow-up
  The patient should indicate satisfaction and relative degree with treatment. All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
Screw malposition rate | 6 months
  Screw malposition rate will be evaluated by a CT scan and the Brantigan score will be applied to document screw fusion.
Incidence of mechanical complications | 2 months, 6 months, 12 months, 24 months and 60 months of follow-up
  Rod Fracture, screw loosening or junctional kyphosis will be evaluated with radiographs
Intraoperative and immediate postoperative outcomes | through study completion, up to 5 years
  Differences in terms of operative time, blood loss, length of stay, time to verticalization, drug use

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Gasbarrini, MD, Principal Investigator — Istituto Ortopedico Rizzoli - Chirurgia vertebrale; Bruna Maccaferri, MD, Study Chair — Istituto Ortopedico Rizzoli -Chirurgia Vertebrale; Francesco Vommaro, MD, Study Chair — Istituto Ortopedico Rizzoli -Chirurgia Vertebrale; Giovanni Ciani, MD, Study Chair — Istituto Ortopedico Rizzoli -Chirurgia Vertebrale; Lucrezia Leggi, MD, Study Chair — Istituto Ortopedico Rizzoli -Chirurgia Vertebrale
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Shakil H, Iqbal ZA, Al-Ghadir AH. Scoliosis: review of types of curves, etiological theories and conservative treatment. J Back Musculoskelet Rehabil. 2014;27(2):111-5. doi: 10.3233/BMR-130438. PMID 24284269
- [Background] Sarwahi V, Horn JJ, Kulkarni PM, Wollowick AL, Lo Y, Gambassi M, Amaral TD. Minimally Invasive Surgery in Patients With Adolescent Idiopathic Scoliosis: Is it Better than the Standard Approach? A 2-Year Follow-up Study. Clin Spine Surg. 2016 Oct;29(8):331-40. doi: 10.1097/BSD.0000000000000106. PMID 24852384
- [Background] Sarwahi V, Galina JM, Hasan S, Atlas A, Ansorge A, De Bodman C, Lo Y, Amaral TD, Dayer R. Minimally Invasive Versus Standard Surgery in Idiopathic Scoliosis Patients: A Comparative Study. Spine (Phila Pa 1976). 2021 Oct 1;46(19):1326-1335. doi: 10.1097/BRS.0000000000004011. PMID 34517401
- [Background] Alhammoud A, Alborno Y, Baco AM, Othman YA, Ogura Y, Steinhaus M, Sheha ED, Qureshi SA. Minimally Invasive Scoliosis Surgery Is a Feasible Option for Management of Idiopathic Scoliosis and Has Equivalent Outcomes to Open Surgery: A Meta-Analysis. Global Spine J. 2022 Apr;12(3):483-492. doi: 10.1177/2192568220988267. Epub 2021 Feb 9. PMID 33557618
- [Background] Neradi D, Kumar V, Kumar S, Sodavarapu P, Goni V, Dhatt SS. Minimally Invasive Surgery versus Open Surgery for Adolescent Idiopathic Scoliosis: A Systematic Review and Meta-Analysis. Asian Spine J. 2022 Apr;16(2):279-289. doi: 10.31616/asj.2020.0605. Epub 2021 May 11. PMID 33966365
- [Background] Si G, Li T, Wang Y, Liu X, Li C, Yu M. Minimally invasive surgery versus standard posterior approach for Lenke Type 1-4 adolescent idiopathic scoliosis: a multicenter, retrospective study. Eur Spine J. 2021 Mar;30(3):706-713. doi: 10.1007/s00586-020-06546-w. Epub 2020 Jul 27. PMID 32720126
- [Derived] Maccaferri B, Filardo G, Cini C, Gasbarrini A, Vommaro F. Adolescent idiopathic scoliosis: a prospective randomised trial protocol comparing clinical and radiological outcomes in minimally invasive surgery versus standard posterior spinal fusion in a single-centre, the Rizzoli Orthopaedic Institute, Bologna, Italy. BMJ Open. 2024 Jul 16;14(7):e075802. doi: 10.1136/bmjopen-2023-075802. PMID 39013643